CLINICAL TRIAL: NCT06967441
Title: Respiratory Virus Infections in Hospitalized Patients With Acute Heart Failure Syndrome: A Prospective Multi-center Observational Study
Brief Title: Respiratory Virus Infections in Acute Heart Failure
Status: Recruiting | Type: Observational
Sponsor: Minjae Yoon (Other)
Collaborators: Samsung Medical Center (Other); Seoul St. Mary's Hospital (Other)
Responsible Party: Sponsor-Investigator, Minjae Yoon, Assistant professor, Seoul National University Bundang Hospital
Organization: Seoul National University Bundang Hospital (Other)
Other Study IDs: SNUBH IRB NO: B-2412-941-302
Record Dates: First submitted 2025-04-17; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Acute Heart Failure Syndrome
Keywords: acute heart failure; respiratory virus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients admitted to the cardiology department with acute heart failure who have a nasopharyngeal respiratory virus PCR test performed within 72 hours of admission will be enrolled in the study cohort.

The detection rate of respiratory viruses including influenza virus, RSV, and coronavirus will be analysed. The investigators will also look for seasonal changes in the frequency of respiratory viruses and differences in the clinical presentation of heart failure based on respiratory virus infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 19 years or older admitted to the cardiology department with acute heart failure
* NT-proBNP >300 pg/mL
* Clinician judgement of possible respiratory viral infection (fever >38 degrees or cough, respiratory symptoms such as sputum or consolidation on x-ray or CRP >5 mg/dL)
* Patients who have a nasopharyngeal swab for respiratory virus PCR test performed within 72 hours of admission for any of the 3 reasons

Exclusion Criteria:

* Patients with a clear other cause of acute heart failure (ex. STEMI, bradycardia requiring a pacemaker, SBP >200mmHg or DBP >110mmHg, haemoglobin <7g/dL)
* If the cause of pulmonary oedema is prominently attributed to exacerbation of CKD
* If there is a clear other source of infection that can explain the fever

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients hospitalised with AHF at three healthcare facilities who had respiratory virus PCR testing performed
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory virus PCR detection rate | Within 3 days of admission
  Respiratory virus PCR detection rate (especially RSV, influenza virus) in acute HF

SECONDARY OUTCOMES:
Days of hospitalization | From admission to discharge during index hospitalization (upto 30 days)
  Days of hospitalization
Rate of ICU care or ventilation | From admission to discharge during index hospitalization (upto 30 days)
  Rate of ICU care or ventilation
In hospital mortality | From admission to discharge during index hospitalization (upto 30 days)
  In hospital mortality
mortality | 12 month
  after discharge, 12-month mortality

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Samsung medical center, Seoul
  - Seoul ST. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No